CLINICAL TRIAL: NCT05553626
Title: Safety and Effectiveness of Left Bundle Branch Pacing (LBBP) in Patients With Cardiac Dysfunction and AV Block
Brief Title: Safety and Effectiveness of Left Bundle Branch Pacing in Patients With Cardiac Dysfunction and AV Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Sir Run Run Shaw Hospital (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shanxi Cardiovascular Hospital (Other); Shanghai 10th People's Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First People's Hospital of Yunnan (Other); Shanghai Zhongshan Hospital (Other); Shenzhen Sun Yat-sen Cardiovascular Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Second Affiliated Hospital of Nanchang University (Other); Tianjin Chest Hospital (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Yan'an Affiliated Hospital of Kunming Medical University (Other); Shanghai Chest Hospital (Other); Medtronic (Shanghai) Management Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FirstWenzhouMU216-02
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-07

CONDITIONS: Atrioventricular Block, Second and Third Degree; Heart Failure; Left Bundle Branch Pacing
Keywords: pacing induced cardiomyopathy; heart failure; pacing; LBBP; BVP; RVP; conduction system pacing; cardiac Resynchronization Therapy; bradycardiac arrhythmia
MeSH Terms: conditions — Atrioventricular Block; Neoplasm Metastasis; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBP Treatment (Experimental): Patients were performed left bundle branch pacing by a single/dual chamber pacemaker or dual chamber ICD device
  Interventions: Device: Left bundle branch pacing; Device: Bi-ventricular pacing
- BVP Treatment (Active Comparator): Patients were performed bi-ventricular pacing by a CRT/CRTD device
  Interventions: Device: Left bundle branch pacing; Device: Bi-ventricular pacing

INTERVENTIONS:
Device: Left bundle branch pacing — Left bundle branch pacing by a single/dual chamber pacemaker or dual chamber ICD device through the pacing lead at left bundle branch region
Device: Bi-ventricular pacing — Bi-ventricular pacing by a CRT/CRTD device

SUMMARY:
This study is a multicenter, prospective, randomized study to assess if cardiac dysfunction patients with LVEF <50% and the estimated ventricular pacing percentage >40% with LBBP have the non-inferior safety and efficacy than CRT on patients' cardiac function and prognosis

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria will be enrolled into the study. In the study, patients with cardiac dysfunction who met the enrollment criteria and will agree to participate in this trial will be 1:1 randomized to the LBBP group and the CRT group. Patients who were successfully implanted were enrolled for evaluation and follow-up. The primary end points of the study is the change of LVEF within 12 months post-implant in both LBBP Treatment Group and CRT Treatment Group

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Agree to participate in trial and sign informed consent
* NYHA cardiac function class I-III
* LVEF<50%
* Second or complete atrioventricular block with pacing indication or ventricular pacing dependent with ventricular pacing percentage >40%
* Patients who are willing to take the de-novo implant or device replacement or upgrade.

Exclusion Criteria:

* Life expectancy <1 year
* Patients with severe tricuspid valvular disease1 or who have undergone mechanical valve or bioprosthetic valve surgery
* Acute myocardial infarction within 1 month
* Women of childbearing age who are pregnant or becoming pregnant during the study period
* Severe liver and kidney dysfunction2
* Have been enrolled in another clinical studies that may interferes with the current trial objectives
* Evidence of severe pulmonary hypertension (PASP>70mmHg)
* Evidence of hypertrophic cardiomyopathy which shall affect the prognosis of patients.
* The investigator believes that subject's physical condition is not suitable for participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change of LVEF | 12 months
  To compare the effects of LBBP Treatment Group and CRT Treatment Group on target subjects by analyzing the LVEF within 12 months post-implant.

SECONDARY OUTCOMES:
Change of LVESV | 12 months
  To demonstrate and compare the LVESV at 12 month post-implant.
successful rate | 12 months
  To characterize the successful rate of LBBP Procedure and CRT Procedure among randomized patients' group.
mortality and heart failure hospitalization rate | 12 months
  To demonstrate and compare the mortality and heart failure hospitalization rate between LBBP and CRT treatment group 12 month post-implant
occurrence of serious complication associated with LBBP procedure | 12 months
  To characterize occurrence of serious complication associated with LBBP procedure within 12 month post-implant.
QRS width between LBBP and CRT | 12 months
  To characterize and compare the QRS width between LBBP and CRT treatment groups during the baseline, preoperative, postoperative and follow up visits within 3 months and 12 month post-implant.
incidence and severity of tricuspid regurgitation | 12 months
  To assess and compare the incidence and severity of tricuspid regurgitation between LBBP and CRT treatment groups within 12 month post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Huang, MD, Principal Investigator — Wenzhou 1st Affliated Hopsital, Wenzhou Medical University
Locations (1):
- First Affliated Hospital, Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No